CLINICAL TRIAL: NCT02334657
Title: Prospective Study of Long-term Outcome After Non-aneurysmal Subarachnoid Hemorrhage
Status: Completed | Type: Observational
Sponsor: University Clinic Frankfurt (Other)
Responsible Party: Principal Investigator, Juergen Konczalla, Dr. med., University Clinic Frankfurt
Other Study IDs: 109/13
Record Dates: First submitted 2015-01-06; First posted 2015-01-08 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Subarachnoid Hemorrhage
Keywords: non-aneurysmal
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- non-aneurysmal subarachnoid hemorrhage: patients with non-aneurysmal subarachnoid hemorrhage, short-term outcome measured by modified Rankin Scale and long-term outcome by SF-36
  Interventions: Other: SF-36
- perimesencephalic SAH: subgroup of non-aneurysmal subarachnoid hemorrhage
  Interventions: Other: SF-36
- non-perimesencephalic (NPM) SAH: subgroup of non-aneurysmal subarachnoid hemorrhage
  Interventions: Other: SF-36
- subgroup of NPM-SAH with Fisher 3: patients with non-aneurysmal (non-perimesencephalic) SAH and a Fisher 3 bleeding pattern
  Interventions: Other: SF-36
- subgroup of NPM-SAH w/o Fisher 3: patients with non-aneurysmal (non-perimesencephalic) SAH and not a Fisher 3 bleeding pattern
  Interventions: Other: SF-36

INTERVENTIONS:
Other: SF-36 — postal questionnaire consisting a short-form health survey with 36 simple questions (SF-36)

SUMMARY:
Spontaneous subarachnoid hemorrhage (SAH) is usually caused by rupture of an intracranial aneurysm, but in up to 15% of patients with spontaneous SAH, no discernible bleeding source can be identified despite of repetitive radiological imaging. Patients, at least 18 months after ictus of a non-aneurysmal SAH, received a regular mail including a letter explaining the study purpose and the postal questionnaire consisting a short-form health survey with 36 simple questions. If we didn't receive answers after three months we made telephone interviews with the patients' family members or their general practitioner.

DETAILED DESCRIPTION:
Spontaneous subarachnoid hemorrhage (SAH) is usually caused by rupture of an intracranial aneurysm, but in up to 15% of patients with spontaneous SAH, no discernible bleeding source can be identified despite of repetitive radiological imaging. The blood distribution can be described as perimesencephalic/prepontine or non-perimesencephalic. Depending on the pattern of SAH the clinical course of the patients can be similar to aneurysmal SAH. In general, patients with a perimesencephalic SAH (PM-SAH) are considered to achieve good outcome and to have lower rebleeding risk. However, long-term outcome data on patients suffering from spontaneous non-aneurysmal SAH (non-aSAH) is scarce and lacking for physical and psychological outcome. Therefore, the aim of the present study was to investigate the long-term physical and psychological outcome in patients suffering from non-aneurysmal spontaneous SAH.

SAH was confirmed on computed tomography (CT) or lumbar puncture. Only patients with a non-traumatic SAH were included. In our hospital algorithm all patients with SAH underwent angiography including 3D digital subtraction angiography (DSA) since 2002 to rule out intracranial sources for SAH. In case of a negative initial angiography, DSA was repeated after 14 days. Additionally, magnetic resonance imaging (MRI) of head/spine was performed to rule out any spinal bleeding sources. In patients with blood distribution exceeding the typical perimesencephalic pattern, a third DSA was performed 3 months after SAH. The first (short-term) follow-up (F/U) was performed six months after ictus. Outcome was measured according to the modified Rankin Scale (mRS) and stratified into favorable (mRS 0-2) and unfavorable (mRS 3-6) after six months. Patients with non-aSAH were divided into perimesencephalic SAH (PM-SAH), non-perimesencephalic SAH (NPM-SAH) and excellent Outcome group (mRS 0). Also the NPM-SAH group was further stratified into Fisher 3 blood pattern and NPM-SAH without Fisher 3 blood pattern.

Patients, at least 18 months after ictus of a non-aneurysmal SAH, received a regular mail including a letter explaining the study purpose and the postal questionnaire consisting a short-form health survey with 36 simple questions. If we didn't receive answers after three months we made telephone interviews with the patients' family members or their general practitioner.

ELIGIBILITY:
Inclusion Criteria:

* spontaneous, non-traumatic SAH
* SAH confirmed on computed tomography (CT) or lumbar puncture
* negative initial and follow-up angiography
* age: no limit

Exclusion Criteria:

* traumatic SAH
* aneurysmal SAH
* SAH in whom other bleeding sources were identified (AVM etc.)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a spontaneous, non-traumatic SAH, in whom no bleeding source was identified by repetitive angiography including 3D digital subtraction angiography
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2013-11; Primary Completion 2014-09 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Long-term outcome of all patients after non-aneurysmal SAH compared to standard population, measured by SF-36 | 18months to 15 years
  Long-term outcome of all patients after non-aneurysmal SAH compared to standard population, measured by SF-36 stratified to:
  * non-aneurysmal SAH
  * PM /NPM-SAH
  * mRS 0 group
  * NPM-SAH: Fisher 3 or non-Fisher 3 bleeding pattern

SECONDARY OUTCOMES:
mortality | 18months to 15 years
  deaths until long-term follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Konczalla, MD, Principal Investigator — Goethe University Hospital, Department of Neurosurgery

REFERENCES:
- [Derived] Konczalla J, Schmitz J, Kashefiolasl S, Senft C, Platz J, Seifert V. Non-aneurysmal non-perimesencephalic subarachnoid hemorrhage: effect of rehabilitation at short-term and in a prospective study of long-term follow-up. Top Stroke Rehabil. 2016 Aug;23(4):261-8. doi: 10.1080/10749357.2016.1149982. Epub 2016 Mar 15. PMID 26916565
- [Derived] Konczalla J, Schmitz J, Kashefiolasl S, Senft C, Seifert V, Platz J. Non-aneurysmal subarachnoid hemorrhage in 173 patients: a prospective study of long-term outcome. Eur J Neurol. 2015 Oct;22(10):1329-36. doi: 10.1111/ene.12762. Epub 2015 Jul 1. PMID 26130053